CLINICAL TRIAL: NCT04609514
Title: Early-phase Studies of a Tailored Evidence-Based Smoking Cessation mHealth App for Persons Living With HIV
Brief Title: Learn to Quit-HIV Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00104423
Record Dates: First submitted 2020-10-22; First posted 2020-10-30 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: HIV/AIDS; Smoking Cessation; Tobacco Use Disorder
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Smoking Cessation; Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Learn to Quit-HIV (Experimental): A smartphone app developed by the research team designed for people with HIV that provides Acceptance and Commitment Therapy skills to address smoking cessation. This app intervention is combined with an 8-week course of nicotine replacement therapy (NRT) patches, along with technical smartphone coaching for the first 4 weeks of the study.
  Interventions: Device: Learn to Quit-HIV; Drug: Nicotine patch; Behavioral: Smartphone coaching
- QuitGuide (Active Comparator): A smartphone app developed by the National Cancer Institute which uses smoking cessation recommendations contained in the US DHHS (United States Department of Health and Human Services) Clinical Practice Guidelines. This app intervention is combined with an 8-week course of nicotine replacement therapy (NRT) patches, along with technical smartphone coaching for the first 4 weeks of the study.
  Interventions: Behavioral: QuitGuide; Drug: Nicotine patch; Behavioral: Smartphone coaching

INTERVENTIONS:
Device: Learn to Quit-HIV — A smartphone app developed by the research team designed for people with HIV that provides Acceptance and Commitment Therapy skills to address smoking cessation.
  Other Names: LTQ-H; LTQ-HIV
  Arms: Learn to Quit-HIV
Behavioral: QuitGuide — A smartphone app developed by the National Cancer Institute which uses smoking cessation recommendations contained in the US DHHS Clinical Practice Guidelines.
  Other Names: NCI QuitGuide
  Arms: QuitGuide
Drug: Nicotine patch — All participants will receive an 8-week course of nicotine patches. They will start off with 4 weeks of 21mg/24 hours patches, then move to 2 weeks of 14mg/24 hours patches, and finally end with 2 weeks of 7mg/24 hours patches.
Behavioral: Smartphone coaching — All participants will partake in over-the-phone smartphone coaching lead by the PI or a research assistant. This will be a time for participants to bring up any technical issues they are experiencing with the study smartphone or app.

SUMMARY:
The study team will conduct a feasibility, acceptability, and preliminary efficacy trial comparing Learn to Quit-HIV (n=30) to an app based on U.S. Clinical Practice Guidelines only (NCI QuitGuide; n=30) among HIV-positive smokers. Both apps will be integrated with NRT and ongoing HIV clinical care.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Currently engaged with an HIV care provider
* Self-report smoking 5 cigarettes or more per day during the past 30 days
* Age 18 years or older
* Current interest in quitting smoking
* Currently own a functioning Android or Apple smartphone

Exclusion Criteria:

* No desire to quit smoking
* Inability to attend study sessions
* Inability to provide informed consent
* Any medical condition or concomitant medication that could compromise subject safety or treatment, as determined by the Principal Investigators and/or Study Physician
* Presence of contraindications for nicotine patch
* Previous allergic reaction or hypersensitivity to nicotine patch (lifetime)
* Current use of nicotine replacement therapy or other smoking cessation treatment (e.g., bupropion, varenicline)
* Pregnant, planning to become pregnant, nursing, or becoming pregnant during the study
* Current untreated and unstable diagnosis of alcohol/substance abuse or dependence (eligible if past abuse/dependence and if receiving treatment and stable for >30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Pacek, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 subjects completed the informed consent process at the screening visit. Eight of these subjects did not pass screen. Therefore, only 43 of these subjects had passed screen and started the study protocol by being assigned to one of the two condition arms.
Groups:
- QuitGuide: A smartphone app developed by the National Cancer Institute which uses smoking cessation recommendations contained in the US DHHS Clinical Practice Guidelines. This app intervention is combined with an 8-week course of nicotine replacement therapy (NRT) patches, along with technical smartphone coaching for the first 4 weeks of the study.
  QuitGuide: A smartphone app developed by the National Cancer Institute which uses smoking cessation recommendations contained in the US DHHS Clinical Practice Guidelines.
  Nicotine patch: All participants will receive an 8-week course of nicotine patches. They will start off with 4 weeks of 21mg/24 hours patches, then move to 2 weeks of 14mg/24 hours patches, and finally end with 2 weeks of 7mg/24 hours patches.
  Smartphone coaching: All participants will partake in over-the-phone smartphone coaching lead by the PI or a research assistant. This will be a time for participants to bring up any technical issues they are experiencing with the study smartphone or app.
Period: Overall Study
Arm/Group | Learn to Quit-HIV | QuitGuide
Started | 22 | 21
Per Protocol Week 4 | 20 | 14
Per Protocol Week 8 | 18 | 12
Per Protocol Week 12 | 15 | 12
Survey or Text Per Protocol Week 12 | 2 | 3
Completed | 17 | 15
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by PI | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Learn to Quit-HIV | QuitGuide | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.59 (11.12) | 52.91 (8.97) | 50.60 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 17 | 14 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 21 | 20 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Duration of Daily App Use
Description: Average duration of app use per arm over participants' 3 months of study participation
Time Frame: 3 months
Population: 7 participants from LTQ arm were excluded from the dataset due to technical/mechanical failure to provide Firebase data. 2 participants were removed from the NCI Quit guide arm due to PI withdrawal.
Measure: Mean (Full Range); unit: minutes
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 15 | 19
minutes | 12 [0 to 260.45] | 1.05 [0 to 472]
Statistical Analysis 1: Comparison: Learn to Quit-HIV vs QuitGuide; Test type: Superiority; p = 0.51, Wilcoxon Rank Sum Test; Median Difference (Final Values) = 10.95

2. Primary Outcome: Frequency of App Use as Measured by Interactions Per Day
Description: Average frequency of app use per arm over participants' 3 months of study participation.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: interactions per day
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 15 | 19
interactions per day | 1.91 (5.30) | 1.21 (5.26)
Statistical Analysis 1: Comparison: Learn to Quit-HIV vs QuitGuide; Test type: Superiority; p < 0.001, Wilcoxon Rank Sum Test

3. Primary Outcome: Participant Attrition at One Month
Description: Number of participants lost to follow-up at one month.
Time Frame: 1 month
Population: Two participants were withdrawn from QuitGuide after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 22 | 19
Participants | 2 | 5

4. Primary Outcome: Participant Attrition at Two Months
Description: Number of participants lost-to-follow-up at two months.
Time Frame: 2 months
Population: Two participants were withdrawn from QuitGuide after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 22 | 19
Participants | 4 | 7

5. Primary Outcome: Participant Attrition at Three Months
Description: Number of participants lost-to-follow-up at three months.
Time Frame: 3 month
Population: Two participants were withdrawn from QuitGuide after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 22 | 19
Participants | 7 | 7

6. Primary Outcome: Recruitment as Measured by the Proportion of Goal Participants Consented
Description: Number of participants consented divided by goal of consenting 60 participants.
Time Frame: 1 year
Population: Target sample size represents the numerator which allows us to calculate the proportion of enrolled participants (n=51) relative to the target goal (N=60). Enrolled participants are those who were consented, however not all consented participants progressed to the next step of study procedure where they would be randomized.
Measure: Number; unit: proportion of goal participants
Groups:
- All Enrolled Participants: Goal of total enrolled participants (n=60) represents the goal of total consents.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 60
proportion of goal participants | 0.85

7. Primary Outcome: App Usability as Measured by the Systems Usability Scale
Description: Average app usability scores as measured by the Systems Usability Scale. The scale has a score range of 0 to 100 with higher scores representing better outcomes.
Time Frame: 1 month or next available time point if participant completed the measure at 3 months.
Population: Two participants from the LTQ arm did not complete the week 4 visit, thus this measure was not obtained. Two participants were withdrawn from Quit Guide after randomization. Three participants from the NCI Quit Guide arm did not complete the week 4 visit, thus this measure was not obtained.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 20 | 14
score on a scale | 73 (16.3) | 78 (15.6)
Statistical Analysis 1: Comparison: Learn to Quit-HIV vs QuitGuide; Test type: Superiority; p = 0.39, Robust Yuen's test — A robust Yuen's test was conducted with an apriori threshold of 0.05 for statistical significance. No covariates were introduced in the model

8. Secondary Outcome: Reduction in Cigarettes Smoked Per Day
Description: Change in cigarettes smoked per day from baseline to the 12-week follow up. Cigarettes smoked per day are measured with a self-report item at baseline and at the 3-month follow up. This outcome is calculated as the difference between cigarettes smoked per day at baseline and the cigarettes smoked per day at the 3 month timepoint. A positive and large values in this outcome indicate larger reductions in cigarettes smoked per day per group, indicating a more positive outcome. A negative and large value indicate an increase in cigarettes smoked per day per group, indicating a clinically negative outcome.
Time Frame: 3 months
Population: Two participants were withdrawn from QuitGuide after randomization. From the LTQ arm, one participant did not complete the measure. From the NCI QuitGuide arm, two participants did not complete the measure and one participant's responses were unusable.
Measure: Mean (Standard Deviation); unit: reduction in cigarettes per day
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 16 | 11
reduction in cigarettes per day | 11.1 (4.91) | 9.2 (5.92)
Statistical Analysis 1: Comparison: Learn to Quit-HIV vs QuitGuide; Test type: Superiority; p = 0.40, Robust Yuen's test

9. Secondary Outcome: Number of Quit Attempts
Description: Quit attempts defined as self-reported no smoking at all for 24 hours; assessed via a Timeline Followback procedure.
Time Frame: 1 month
Population: Participants who completed a Timeline Followback were included in the analysis.
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 9 | 10
quit attempts | 1.89 (1.45) | 1.30 (0.82)
Statistical Analysis 1: Comparison: Learn to Quit-HIV vs QuitGuide; Test type: Superiority; p = 0.478, Wilcoxon rank sum test; Wilcoxon rank sum test with continuity correction

10. Secondary Outcome: Number of Quit Attempts
Description: Quit attempts defined as self-reported no smoking at all for 24 hours; assessed via a Timeline Followback procedure.
Time Frame: 3 months
Population: Participants who completed a Timeline Followback were included in the analysis.
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 7 | 6
quit attempts | 1.86 (1.68) | 2.50 (1.38)
Statistical Analysis 1: Comparison: Learn to Quit-HIV vs QuitGuide; Test type: Superiority; p = 0.51, Wilcoxon rank sum test; Wilcoxon rank sum test with continuity correction

11. Secondary Outcome: 7-day Point Prevalence Abstinence
Description: Percent of subjects in each group reporting 7-day point prevalence abstinence. Abstinence is determined by a self-report of not smoking any tobacco product at all during the corresponding time frame period, AND by a result of less than 5 ppm in carbon monoxide breath testing. If the participant does not meet both criteria, or if they do not provide data at the time-point they are not considered abstinent.
Time Frame: 1 month
Population: Data not collected.
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: 7-day Point Prevalence Abstinence
Description: as for outcome 11
Time Frame: 3 months
Population: The Intention to Treat sample was utilized for this outcome. Two participants were withdrawn from QuitGuide after randomization. Lost to follow up participants were assumed to have maintained their smoking status.
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 22 | 19
percentage of participants | 18.2 (0.395) | 15.8 (0.375)
Statistical Analysis 1: Comparison: Learn to Quit-HIV vs QuitGuide; Test type: Superiority; p = 0.8392, Regression, Logistic; Odds Ratio (OR) = 1.185, 95% CI 2-sided [0.23 to 6.119]

13. Secondary Outcome: Overall Adherence to Nicotine Replacement Therapy
Description: Reported as percent of participants who used the patch at least 80% of the days of the required 8 weeks. Adherence determined by timeline follow back interview.
Time Frame: baseline to 3 months
Population: Two participants from LTQ arm did not complete the measure. Two participants were withdrawn from QuitGuide after randomization. Four participants from QuitGuide arm did not complete the measure.
Measure: Number; unit: percentage of participants
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 20 | 15
percentage of participants | 31.8 | 31.6
Statistical Analysis 1: Comparison: Learn to Quit-HIV vs QuitGuide; Test type: Superiority; p = 1.00, Pearson's Chi-squared test; Pearson's Chi-squared test with Yates' continuity correction

14. Secondary Outcome: Number of Participants With at Least One Adverse Event Determined to be Related to the Study Interventions
Description: Adverse events reported here will only include those that are determined to be related to the study interventions.
Time Frame: 3 months
Population: Two participants were withdrawn from QuitGuide after randomization. All participants who were randomized were included in the analysis as total population that could have reported adverse events related to the study during their enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit-HIV | QuitGuide
Number analyzed (Participants) | 22 | 19
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Learn to Quit-HIV | QuitGuide
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 6/22 | 5/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Learn to Quit-HIV (N=22) | QuitGuide (N=21)
Cough (Infections and infestations) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COVID (Infections and infestations) | 1 | 1
Diabetes Diagnosis (Endocrine disorders) | 1 | 0
Infection (dermis) (Infections and infestations) | 1 | 0
Muscle Ache (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Sweating (Skin and subcutaneous tissue disorders) | 1 | 0
COPD Diagnosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Headache (General disorders) | 0 | 1
Muscle Pain (Injury, poisoning and procedural complications) | 0 | 1
Nasal congestion (Infections and infestations) | 0 | 1
Numbness/Tingling (Nervous system disorders) | 0 | 1
Procedure (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT04609514/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT04609514/ICF_000.pdf